CLINICAL TRIAL: NCT05976945
Title: Imagery Rescripting as a Stand-alone Treatment for Depression: a Pilot Study.
Brief Title: Imagery Rescripting as Treatment for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Collaborators: Academic Center for Trauma and Personality (Unknown)
Responsible Party: Principal Investigator, Arnoud Arntz, Professor, University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-CP-14288
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Persistent Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Multiple baseline case series design: by randomizing participants to different lengths of waitlist (baseline) and comparing means and slopes of weekly reported depression severity and core beliefs, the effectiveness of the treatment is tested.
Masking Description: The investigator will not have access to assignment of participants to waitlist length and the data until data collection is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline-Preparation-Imagery Rescripting-Post Treatment (Experimental): Each participant follows this sequence: (1) 6-10 weeks waitlist during which no treatment is offered; (2) 5 weekly preparatory sessions. During these sessions the rationale of ImRs will be explained in more detail and a list of painful (childhood) memories to be addressed with ImRs is to be compiled, based on any further input from the patient; and a case conceptualization is made; (3) 8 to 12 sessions (45-60 minutes) of ImRs will be offered to participating patients. The stand-alone ImRs treatment will be based upon the protocol described by Arntz & Weertman (1999). (This protocol can be modified to tailor the needs of this study more specifically. Possible adaptations shall be based upon the manual developed by Brewin and colleagues (2009) for their study of applying ImRs to depression.); (4) After end of active treatment (ImRs) 5 weeks follow during which only weekly assessments are done.
  Interventions: Behavioral: Imagery Rescripting

INTERVENTIONS:
Behavioral: Imagery Rescripting — In Imagery Rescripting patients imagine a different sequence of events matching their needs better than what actually happened in traumatic and other adverse (childhood) experiences.

SUMMARY:
The goal of this multiple baseline case series study is to test Imagery Rescripting in depression. The main question[s] it aims to answer are:

* does Imagery Rescripting lead to a reduction of depression and of believability of negative beliefs held by the participants?
* does Imagery Rescripting also leads to reductions in worrying and brooding?
* Participants will wait for 6-10 weeks (to assess time effects without treatment), followed by 5 weekly preparation sessions, 8-12 weekly Imagery Rescripting sessions, and 5 weeks post-treatment.
* Participants will rate the believability of 3-5 core dysfunctional beliefs related to their depression as well as 2 items assessing depression severity on a weekly basis. In addition, they will fill out more extensive questionnaires on depression, worry and brooding before each phase, as well as at 5 weeks post-treatment, and 6 and 12 months follow-up.

DETAILED DESCRIPTION:
In a multiple baseline case series study the effectiveness of Imagery Rescripting (ImRs) as a treatment for depression will be tested. 10 patients with a major depressive disorder (MDD) or a persistent depressive disorder (PDD) will be randomized to different waitlist lengths (6-10 weeks), after which they will enter a 5-session preparation phase (5 weeks), followed by 12 weekly sessions of ImRs. After this treatment follow-up assessments take place at 5 weeks, 6 and 12 months. Primary outcomes are (1) depression severity weekly assessed with the Patient Health Questionnaire (PHQ-2) and (2) idiosyncratic core beliefs assessed with visual analogue scales. The hypothesis is that primary outcomes reduce more during treatment than during wait or preparation and remain stable or further improve post-treatment. Similarly, for secondary outcomes (depression severity assessed with the Beck Depression Inventory II (BDI-II); brooding (dysfunctional type of rumination) assessed with the Ruminative Response Scale (RRS) Brooding subscale; and worrying assessed with the Penn State Worry Questionnaire (PSWQ)) we expect the largest improvement to take place from pre- to post treatment, with little change taking place during baseline and preparation, and during/after post-treatment.

Results will be analyzed by multilevel analysis, pooling the effects of the individual cases. Lastly, participants will be interviewed 5 weeks post treatment about their experiences with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of MDD as assessed with the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) (SCID-5)
* Total score of 20* or above on the BDI-II (cut-off score for moderate depression) (Beck et al., 1996). (*Based on previous research by Brewin et al. (2009) & Yuen-tin (2017) demonstrating averages of BDI-II: 34-35, in their population.)
* Age 18-65
* Dutch or English as a first language (or estimated as sufficient to receive treatment in either of these languages without interpreter)
* Willingness to participate in the study (signed informed consent)

Exclusion Criteria:

* DSM-5 Bipolar disorder, type 1 (current or past); if there has been no manic episode the last year patients will be included
* Psychotic disorders (though psychotic features alongside depression will be allowed)
* Organic brain disease
* Intelligence Quotient (IQ) < 80
* High risk of self-harm or suicide
* Current substance abuse severe level
* Start of new medication within 2 months before beginning the study (medication used for longer periods can be continued; patients are requested to keep medication stable during the course of the study)
* Having received ImRs (either as a stand-alone or embedded in a greater treatment such as cognitive behavior therapy (CBT) or schema therapy) within the last year
* No other evidence-based treatment of MDD is allowed during the study.
* Not able to plan enough time for weekly therapy sessions (45-60 minutes); weekly measurements (estimate of 5 minutes) and other measurements (estimate of 20 minutes); and the qualitative post-treatment interview (estimate of 60 minutes) during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Depression severity | 28-32 weeks plus 6 and 12 months follow-ups
  Depression severity assessed with the first 2 items of the Patient Health Questionnaire-9. The minimum score is 0, the maximum score is 6. A higher score means worse outcome.
Core beliefs strength | 28-32 weeks plus 6 and 12 months follow-ups
  Idiosyncratic core beliefs related to the depression are formulated together with the participant and weekly rated on Visual Analogue Scales.The mean of the scores is taken, range 0-100. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Beck Depression Inventory-II | before baseline, before preparatory sessions, before ImRs treatment, 5 weeks after ImRs treatment, 6 and 12 months follow-ups
  The Beck Depression Inventory-II assesses severity of depression. The minimum score is 0, the maximum score is 63. Higher scores mean worse outcomes.
Brooding intensity | before baseline, before preparatory sessions, before ImRs treatment, 5 weeks after ImRs treatment, 6 and 12 months follow-ups
  The Brooding subscale of the Ruminative Response Scale assesses intensity of problematic brooding. The minimum score is 5, the maximum is 20. Higher scores mean worse outcomes.
Worry intensity | before baseline, before preparatory sessions, before ImRs treatment, 5 weeks after ImRs treatment, 6 and 12 months follow-ups
  The Penn State Worry Questionnaire assesses intensity of problematic worrying. The minimum score is 16, the maximum 80. Higher scores mean worse outcomes.

OTHER OUTCOMES:
patients' experiences | 5 weeks after end of treatment
  with a semi-structured interview, participants will be interviewed 5 weeks after treatment. A qualitative analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Arnoud Arntz, PhD, Principal Investigator — University of Amsterdam
Locations (1):
- Academic Center for Trauma and Personality ACTP, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
because of privacy regulations individual patient data cannot be shared, unless the European Union (EU) regulations on data protection are guaranteed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT05976945/Prot_SAP_000.pdf